CLINICAL TRIAL: NCT04541914
Title: Diagnostic Efficacy of Peripheral Blood Marker-based Molecular Diagnostic Method for Antibody-mediated Rejection (AMR) in ABO Blood Type Incompatible Kidney Transplant (ABOiKT)
Brief Title: Diagnostic Efficacy of Molecular Diagnostic Method for AMR in ABOiKT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Jaeseok Yang, Principal Investigator, Seoul National University Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 20030871109
Record Dates: First submitted 2020-08-27; First posted 2020-09-09 (Actual); Last update posted 2025-05-15 (Actual); Status verified 2024-04

CONDITIONS: ABO Blood Type Incompatible Kidney Transplantation; Antibody-mediated Rejection
Keywords: molecular diagnostic method; diagnostic efficacy; accommodation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Validation group (Experimental): Evaluation for diagnostic efficacy of peripheral blood marker-based molecular diagnostic method for antibody-mediated rejection (AMR) in ABO blood type incompatible kidney transplant (ABOiKT)
  Interventions: Diagnostic Test: 5-gene classification model

INTERVENTIONS:
Diagnostic Test: 5-gene classification model — Peripheral blood marker-based molecular diagnostic method for AMR in ABOiKT

SUMMARY:
The purpose of this study is to determine whether the peripheral blood marker-based molecular diagnostic method developed in the previous study can differentiate and predict accommodation and antibody-mediated rejection (AMR) in ABO blood type incompatible kidney transplant (ABOiKT) patients who are prospectively recruited.

DETAILED DESCRIPTION:
Our research team retrospectively analyzes biomarkers that distinguish accommodation and acute antibody-mediated rejection through transcriptomic analysis of peripheral blood in patients with ABO blood type incompatibility kidney transplantation at Seoul National University Hospital. Through this, a classification model was developed to distinguish accommodation and antibody-mediated rejection using peripheral blood marker at the time of the protocol biopsy on the 10th day after renal transplantation, and recently reported as a new peripheral blood marker-based molecular diagnostic method. On the 10th day after surgery, transcriptomic analysis through RNA-seq was performed using samples of peripheral blood from 18 patients with accommodation and 10 patients with antibody-mediated rejection confirmed by protocol biopsy. The candidate genes were validated in the discovery set and another independent training set through quantitative real-time polymerase chain reaction (PCR). Finally, a 5-gene classification model including COX7A2L, CD69, CD14, CFD, and FOXJ3 was developed through logistic regression analysis.

To evaluate the diagnostic effectiveness (sensitivity, specificity) for the peripheral blood marker-based molecular diagnostic method by prospectively recruiting patients with ABO blood type incompatible kidney transplantation is needed. And, it is necessary to evaluate the effectiveness of whether the peripheral blood marker-based molecular diagnostic method can predict antibody-mediated rejection or accommodation as a result of protocol biopsy that will be performed on the 10th day after transplantation - peripheral blood samples collected earlier than the 10th day (day 5 and day 7) after ABO blood type incompatible kidney transplantation.

ELIGIBILITY:
Inclusion Criteria:

* ABO blood group incompatible kidney transplant patients
* Patients who consent to written consent
* Patients over 19 years of age

Exclusion Criteria:

* Pregnant patients
* Patients with a history of drug abuse within the last 6 months
* Psychiatric disease history (major depression, bipolar disorder, schizophrenia, etc.)
* Patients who do not want to participate in this study

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2020-05-19 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2023-12-31 (Actual)

PRIMARY OUTCOMES:
The value by logistic regression equation using peripheral blood marker on the 7th day after ABOiKT for prediction of antibody-mediated rejection | the 7th day after ABO-incompatible kidney transplantation
  To evaluate whether the value by logistic regression equation using peripheral blood marker-based molecular diagnostic method on the 7th day after ABOiKT can predict antibody-mediated rejection from the protocol kidney biopsy results on the 10±2 day after ABOiKT (If the probability value of a sample is higher than 0.5, it is classified as accommodation. Samples with values <0.5 are classified as antibody-mediated rejection by this diagnostic method)

SECONDARY OUTCOMES:
The value by logistic regression equation using peripheral blood marker on the 5th or 10th day after ABOiKT for prediction of antibody-mediated rejection | the 5th or 10th day after ABO-incompatible kidney transplantation
  To evaluate whether the value by logistic regression equation using peripheral blood marker-based molecular diagnostic method on the 5th or 10th day after ABOiKT can predict antibody-mediated rejection from the protocol kidney biopsy results on the 10±2 day after ABOiKT (If the probability value of a sample is higher than 0.5, it is classified as accommodation. Samples with values <0.5 are classified as antibody-mediated rejection by this diagnostic method)

CONTACTS AND LOCATIONS:
Overall Officials: Jaeseok Yang, M.D., Ph.D, Principal Investigator — Transplantation Center, Seoul National University Hospital
Locations (1):
- Seoul National University Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Jeon HJ, Lee JG, Kim K, Jang JY, Han SW, Choi J, Ryu JH, Koo TY, Jeong JC, Lee JW, Ishida H, Park JB, Lee SH, Ahn C, Yang J. Peripheral blood transcriptome analysis and development of classification model for diagnosing antibody-mediated rejection vs accommodation in ABO-incompatible kidney transplant. Am J Transplant. 2020 Jan;20(1):112-124. doi: 10.1111/ajt.15553. Epub 2019 Aug 26. PMID 31373158